CLINICAL TRIAL: NCT06441214
Title: Retrospective-prospective Study to Evaluate Treatment Management and Outcomes of Patients With Waldenström's Macroglobulinemia (WM) Treated in Italy According to the Zanubrutinib (Brukinsa®) Compassionate Use Program (CUP) and in Common Practice Following Commercial Approval
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Other Study IDs: FIL_BRUCE-ITA
Record Dates: First submitted 2024-05-15; First posted 2024-06-04 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Waldenström's Macroglobulinemia (WM)
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — zanubrutinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: All patients with Waldenström's macroglobulinemia enrolled in Pre-Reimbursement Access Program (PRAP) of Zanubrutinib, as per Compassionate Use Program (CUP) of Zanubrutinib, and patients treated with commercial drug (Brukinsa®) from PRAP closure to the study start.
- Prospective cohort: Patients with Waldenström's macroglobulinemia treated with Zanubrutinibin clinical practice enrolled from the study start up to 12 months.
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — Patients will be treated with Zanubrutinib as per routine clinical practice.
  Groups: Prospective cohort

SUMMARY:
This is a non-interventional, observational, retrospective and prospective multicenter Italian study, to describe treatment management and outcomes of Waldenström's Macroglobulinemia (WM) patients treated according to the Italian Compassionate Use Program (CUP) and receiving zanubrutinib following its commercial approval.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form
* Waldenström's macroglobulinemia diagnosis in need of treatment according to ESMO (European Society for Medical Oncology) guideline 2018
* Patients who received Zanubrutinib according to the Italian CUP or in common practice following Zanubrutinib commercial approval
* Treatment with zanubrutinib according to current SmPC (Summary of Product Characteristics)
* Treatment decision before inclusion into this non-interventional study
* Age ≥18 years

Exclusion Criteria:

* Contraindications according to SmPC for patients with WM
* Participation in an interventional clinical trial during zanubrutinib treatment
* Patients with disease progression during a BTKi treatment (if pre-treated with BTK, only those intolerants are considered eligible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Waldenström's Macroglobulinemia (WM) treated in Italy according to the Zanubrutinib (Brukinsa®) compassionate use program (CUP) and in common practice following commercial approval.
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2024-12-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of treatment discontinuation due to toxicity | From the date of first zanubrutinib administration to the date of definitive treatment discontinuation or dose reduction for any cause or death from any cause, from october 2020 up to 24 months since study start
  Cumulative incidence of treatment discontinuation due to toxicity

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Retrospective cohort: from october 2020 until the study start. Prospective cohort: up to 24 months (duration of study)
  Incidence of adverse events (AEs)
Incidence of adverse events related to zanubrutinib. | Retrospective cohort: from october 2020 until the study start. Prospective cohort: up to 24 months (duration of study)
  Incidence of adverse events related to zanubrutinib.
Incidence of relevant adverse events. | Retrospective cohort: from october 2020 until the study start. Prospective cohort: up to 24 months (duration of study)
  Incidence of relevant adverse events.
Incidence of serious adverse events (SAEs). | Retrospective cohort: from october 2020 until the study start. Prospective cohort: up to 24 months (duration of study)
  Incidence of serious adverse events (SAEs).
Incidence of adverse events leading to death. | Retrospective cohort: from october 2020 until the study start. Prospective cohort: up to 24 months (duration of study)
  Incidence of adverse events leading to death.
Incidence of adverse events leading to treatment discontinuation. | Retrospective cohort: from october 2020 until the study start. Prospective cohort: up to 24 months (duration of study)
  Incidence of adverse events leading to treatment discontinuation.
Incidence of adverse events leading to dose reduction/interruption. | Retrospective cohort: from october 2020 until the study start. Prospective cohort: up to 24 months (duration of study)
  Incidence of adverse events leading to dose reduction/interruption.
Time to first onset of relevant adverse event. | Retrospective cohort: from october 2020 until the study start. Prospective cohort: up to 24 months (duration of study)
  Time to first onset of relevant adverse event.
AEs ≥ G3 Hematological and non-hematological. | Retrospective cohort: from october 2020 until the study start. Prospective cohort: up to 24 months (duration of study)
  AEs ≥ G3 Hematological and non-hematological.
Impact of patients' characteristics and comorbidities on G3 or higher AEs and relevant adverse events development. | Retrospective cohort: from october 2020 until the study start. Prospective cohort: up to 24 months (duration of study)
  Impact of patients' characteristics and comorbidities on G3 or higher AEs and relevant adverse events development.
Frequency of transformation of WM to an aggressive lymphoma and frequency of secondary malignancies. | Retrospective cohort: from october 2020 until the study start. Prospective cohort: up to 24 months (duration of study)
  Frequency of transformation of WM to an aggressive lymphoma and frequency of secondary malignancies.
Major response rate (MRR) | Retrospective cohort: from october 2020 until the study start. Prospective cohort: up to 24 months (duration of study)
  Major response rate (MRR) (≥PR) (best reported response).
Overall response rate (ORR) | Retrospective cohort: from october 2020 until the study start. Prospective cohort: up to 24 months (duration of study)
  Overall response rate (ORR, defined as MRR plus minor response rate)
Best response | Retrospective cohort: from october 2020 until the study start. Prospective cohort: up to 24 months (duration of study)
  Best response (best reported response).
Progression-free survival (PFS) | Retrospective cohort: from october 2020 until the study start. Prospective cohort: up to 24 months (duration of study)
  Progression-free survival (PFS) including 6, 12, and 24-month PFS rate
Overall survival (OS) | Retrospective cohort: from october 2020 until the study start. Prospective cohort: up to 24 months (duration of study)
  Overall survival (OS) including 6, 12, and 24-month OS rate.
Time to treatment failure | Retrospective cohort: from october 2020 until the study start. Prospective cohort: up to 24 months (duration of study)
  Time to treatment failure (any treatment definitive discontinuation, incl. patient or investigator decision, toxicity, progression or death).
Duration of response (DOR) | Retrospective cohort: from october 2020 until the study start. Prospective cohort: up to 24 months (duration of study)
  Duration of response (DOR)
Change of IgM levels until end of zanubrutinib treatment. | Retrospective cohort: from october 2020 until the study start. Prospective cohort: up to 24 months (duration of study)
  Change of IgM levels until end of zanubrutinib treatment.
Impact of patients and disease characteristics, and biomarker test results (MYD88 and CXCR4, if available) on treatment response. | Retrospective cohort: from october 2020 until the study start. Prospective cohort: up to 24 months (duration of study)
  Impact of patients and disease characteristics, and biomarker test results (MYD88 and CXCR4, if available) on treatment response.
Hospital stays | Retrospective cohort: from october 2020 until the study start. Prospective cohort: up to 24 months (duration of study)
  Hospital stays comprises all planned and unplanned hospitalizations as well as emergency unit visits, regardless of whether there is an association with WM or not. All hospitalizations and emergency unit visits that started during therapy with zanubrutinib will be considered for hospital stays.
EORTC-QLQ-C30 | Prospective cohort: up to 24 months (duration of study)
  Quality of life (QoL) assessed with EORTC-QLQ-C30 questionnaire
EQ-5D-5L | Prospective cohort: up to 24 months (duration of study)
  Quality of life (QoL) assessed with EQ-5D-5L questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria Frustaci, Principal Investigator — ASST Grande Ospedale Metropolitano Niguarda, Milano, Italy
Locations (28):
- Italy (28):
  - A.O. SS. Antonio e Biagio e Cesare Arrigo - S.C.D.U. Ematologia, Alessandria
  - A.O.U. Ospedali Riuniti - Clinica di Ematologia, Ancona
  - Ospedale C. e G. Mazzoni - U.O.C. di Ematologia, Ascoli Piceno
  - AOU Policlinico Consorziale - U.O. Ematologia con Trapianto, Bari
  - Nuovo Ospedale degli Infermi - SSD Ematologia, Biella
  - Policlinico S. Orsola-Malpighi - Istituto di Ematologia "Seragnoli", Bologna
  - Ospedale Centrale di Bolzano - Divisione di Ematologia e T.M.O., Bolzano
  - Azienda Ospedaliera Universitaria Policlinico - S. Marco - UOC di Ematologia, Catania
  - Azienda Ospedaliero-Universitaria di Ferrara - Arcispedale Sant'Anna - Ematologia e fisiopatologia della coagulazione, Ferrara
  - Azienda Ospedaliera Universitaria Careggi - Unità funzionale di Ematologia, Florence
  - Ospedale Policlinico San Martino S.S.R.L. - IRCCS per l'Oncologia - Ematologia e terapie cellulari, Genova
  - ASST Grande Ospedale Metropolitano Niguarda - S.C. Ematologia, Milan
  - IEO Istituto Europeo di Oncologia - Divisione Ematoncologia, Milan
  - Ospedale Maggiore Policlinico - Fondazione IRCCS Ca Granda - Ematologia, Milan
  - AOU Maggiore della Carità di Novara - SCDU Ematologia, Novara
  - AOU di Padova - Ematologia, Padua
  - A.O. Ospedali Riuniti Villa Sofia-Cervello - Divisione di Ematologia, Palermo
  - RCCS Policlinico S. Matteo di Pavia - Div. di Ematologia, Pavia
  - P.O. Spirito Santo di Pescara - UOC Ematologia Dipartimento Oncologico Ematologico - ASL Pescara, Pescara
  - AOU Pisana - U.O. Ematologia, Pisa
  - Ospedale delle Croci - Ematologia, Ravenna
  - Azienda Unità Sanitaria Locale-IRCCS - Arcispedale Santa Maria Nuova - Ematologia, Reggio Emilia
  - Università Cattolica Sacro Cuore - Ematologia, Roma
  - AOU Senese - U.O.C. Ematologia, Siena
  - Ospedale "G. Mazzini" - UOS Ematologia, Teramo
  - A.O.U. Città della Salute e della Scienza di Torino - Ematologia Universitaria, Torino
  - A.O.U. Città della Salute e della Scienza di Torino - S.C. Ematologia, Torino
  - Azienda Sanitaria Universitaria Friuli Centrale (ASU FC) - SOC Clinica Ematologica, Udine